CLINICAL TRIAL: NCT00324116
Title: A Prospective, Open-Label Multi Center Trial Evaluating The Safety And Efficacy Of 0.3 Mg/Eye Pegaptanib Sodium (Macugen) Intravitreous Injection Given Every 6 Weeks For 54 Weeks In Patients With Small Neovascular Age-Related Macular Degeneration (AMD) Lesions
Brief Title: Evaluation Of Safety And Efficacy Of 0.3 Mg/Eye Macugen In Patients With Small Age-Related Macular Degeneration Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: ITEC GROUP 3 (Unknown)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5751016
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2010-03

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental)
  Interventions: Drug: pegaptanib sodium (Macugen)

INTERVENTIONS:
Drug: pegaptanib sodium (Macugen) — 0.3 MG/eye pegaptanib IB sodium by intravitreous injection given every 6 weeks for 54 weeks.
  Other Names: MACUGEN

SUMMARY:
To evaluate the efficacy, based on the best-corrected visual acuity (using the ETDRS chart), of a 0.3 mg/eye pegaptanib sodium intravitreous injection given every 6 weeks for 54 weeks in patients with exudative age-related macular degeneration and evidence of recent onset, subfoveal and/or juxtafoveal choroidal neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and angiographic evidence of juxtafoveal or subfoveal choroidal neovascularization secondary to AMD with a total lesion size of less than 2 MPS disc areas
* Best-corrected visual acuity in the study eye greater than 54 letters (ETDRS)
* Women must be using 2 forms of effective contraception
* Adequate hematological, renal and liver functions

Exclusion Criteria:

* Any atrophy or fibrosis; any retinal hemorrhage measuring more than 1 disc area
* Any extrafoveal choroidal neovascularization
* Any intraocular surgery or thermal laser to the study eye within 3 months of enrollment
* Previous or concomitant therapy for AMD including PDT with verteporfin (Visudyne) or subfoveal/non-foveal thermal laser therapy, transpupillary thermotherapy, external beam radiation, submacular surgery.
* Presence of other causes of choroidal neovascularization, including pathological myopia, the ocular histoplasmosis syndrome, angioid streaks, choroidal rupture and multifocal choroiditis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- France (27):
  - Pfizer Investigational Site, Angers, Cedex 09
  - Pfizer Investigational Site, Lyon, Cedex 4
  - Pfizer Investigational Site, Besançon, Cedex
  - Pfizer Investigational Site, Créteil, Cedex
  - Pfizer Investigational Site, Mâcon, Cedex
  - Pfizer Investigational Site, Poitiers, Cedex
  - Pfizer Investigational Site, Bayonne
  - Pfizer Investigational Site, Belfort
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, La Rochefoucauld
  - Pfizer Investigational Site, La Tronche
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rives
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Herblain
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751016&StudyName=Evaluation%20Of%20Safety%20And%20Efficacy%20Of%200.3%20Mg/Eye%20Macugen%20In%20Patients%20With%20Small%20Age-Related%20Macular%20Degeneration%20Lesions

RESULTS

PARTICIPANT FLOW:
Groups:
- Pegaptanib Sodium: All subjects received a 0.3 mg/eye pegaptanib sodium intravitreous injection every 6 weeks for 54 weeks.
Period: Overall Study
Arm/Group | Pegaptanib Sodium
Started | 81 (subjects received treatment)
Completed | 49
Not Completed | 32
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 17
Not completed — Withdrawal by Subject | 5
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 81
Age Continuous [Mean (Standard Deviation); unit: years] | 76.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders for Visual Acuity Using Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: Best-corrected visual acuity assessed using retroilluminated modified Ferris-Bailey ETDRS charts. When possible to measure visual acuity @ 2.0 m (≥20 letters), visual acuity score for that eye recorded as number of letters correct plus 15; otherwise, score was number of letters read correctly @ 1.0 m plus number, if any, read @ 2.0 m. If no letter was read correctly either at 2.0 or 1.0 m, then visual acuity score was recorded as 0. Responders defined as subjects having lost from baseline less than 15 letters of the best-corrected visual acuity; includes subjects with visual acuity gain.
Time Frame: Baseline, 54 Weeks
Population: The full analysis set (FAS) was derived from the set of all enrolled subjects who 1) were administered the study medication AND 2) had post-baseline documentation of efficacy available. In the case of missing data post-baseline, the subject was considered censored at the time of the last available data for the score.
Measure: Number; unit: participants
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
participants
  Responders | 40 [76 to 95]
  Non-Responders | 7
  Censored (subjects with missing data) | 33
Statistical Analysis 1: Comparison: Pegaptanib Sodium; Test type: Superiority or Other; percent responders = 85, 95% CI [76 to 95] — Proportion of responders estimated by Kaplan-Meier analysis. Proportion of responders along with 95% CI calculated directly from estimate of survival distribution function. Percentage denominator = total number of subjects without missing data

2. Secondary Outcome: Change From Baseline in Visual Acuity
Description: Best-corrected visual acuity assessed using retroilluminated modified Ferris-Bailey ETDRS charts. When possible to measure visual acuity @ 2.0 m (≥20 letters), visual acuity score for that eye recorded as number of letters correct plus 15; otherwise, score was number of letters read correctly @ 1.0 m plus number, if any, read @ 2.0 m. If no letter was read correctly either at 2.0 or 1.0 m, then visual acuity score was recorded as 0. Change: mean score at observation minus mean score at baseline.
Time Frame: Baseline, 6 weeks, 12 weeks, 54 weeks
Population: FAS; n=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
score on scale
  6 weeks (n=76) | -4.29 (11.11)
  12 weeks (n=74) | -5.86 (13.79)
  54 weeks (n=49) | -11.12 (17.96)
Statistical Analysis 1: Comparison: Pegaptanib Sodium; 6 weeks; Test type: Superiority or Other; Mean Difference (Net) = -4.29, 95% CI [-6.83 to -1.75] — 95% CI for the change in mean value obtained from one sample t-test
Statistical Analysis 2: Comparison: Pegaptanib Sodium; 12 weeks; Test type: Superiority or Other; Mean Difference (Net) = -5.86, 95% CI [-9.06 to -2.67] — 95% CI for the change in mean value obtained from one sample t-test
Statistical Analysis 3: Comparison: Pegaptanib Sodium; 54 weeks; Test type: Superiority or Other; Mean Difference (Net) = -11.12, 95% CI [-16.28 to -5.96] — 95% CI for the change in mean value obtained from one sample t-test

3. Secondary Outcome: Number of Subjects Gaining Vision
Description: Subjects gaining vision: gain from baseline of more than 15 letters of visual acuity. Best-corrected visual acuity assessed using retroilluminated modified Ferris-Bailey ETDRS charts. When possible to measure visual acuity @ 2.0 m (≥20 letters), visual acuity score for that eye recorded as number of letters correct plus 15; otherwise, score was number of letters read correctly @ 1.0 m plus number, if any, read @ 2.0 m. If no letter was read correctly either at 2.0 or 1.0 m, then visual acuity score was recorded as 0.
Time Frame: 54 weeks or at early termination
Population: FAS
Measure: Number; unit: participant
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
participant
  Gained | 4
  Did not gain | 74
  Assessment Not Done | 2
Statistical Analysis 1: Comparison: Pegaptanib Sodium; Test type: Superiority or Other; percentage of subjects = 5.00, 95% CI [1.61 to 11.32] — Proportion of subjects gaining vision was estimated on an observed case basis. Percentage denominator = total number of subjects in the FAS. 95% confidence intervals were calculated from Fleiss quadratic equations

4. Secondary Outcome: Number of Subjects Maintaining Vision
Description: Subjects maintaining vision: gain from baseline of more than 0 letters of visual acuity. Best-corrected visual acuity assessed using retroilluminated modified Ferris-Bailey ETDRS charts. When possible to measure visual acuity @ 2.0 m (≥20 letters), visual acuity score for that eye recorded as number of letters correct plus 15; otherwise, score was number of letters read correctly @ 1.0 m plus number, if any, read @ 2.0 m. If no letter was read correctly either at 2.0 or 1.0 m, then visual acuity score was recorded as 0.
Time Frame: 54 weeks or at early termination
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
participants
  Maintained | 18
  Did not maintain | 60
  Not Done | 2
Statistical Analysis 1: Comparison: Pegaptanib Sodium; Test type: Superiority or Other; percentage of subjects = 22.50, 95% CI [14.22 to 32.11] — Proportion of subjects maintaining vision was estimated on an observed case basis. Percentage denominator = total number of subjects in the FAS. 95% confidence intervals were calculated from Fleiss quadratic equations

5. Secondary Outcome: Number of Subjects With Severe Visual Loss
Description: Subjects with severe visual loss: loss from baseline of >= 30 letters of visual acuity. Best-corrected visual acuity assessed using retroilluminated modified Ferris-Bailey ETDRS charts. When possible to measure visual acuity @ 2.0 m (≥20 letters), visual acuity score for that eye recorded as number of letters correct plus 15; otherwise, score was number of letters read correctly @ 1.0 m plus number, if any, read @ 2.0 m. If no letter was read correctly either at 2.0 or 1.0 m, then visual acuity score was recorded as 0.
Time Frame: 54 weeks or at early termination
Population: FAS
Measure: Number; unit: participants
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
participants
  Severe Loss | 11
  Not severe loss | 67
  Not Done | 2
Statistical Analysis 1: Comparison: Pegaptanib Sodium; Test type: Superiority or Other; percentage of subjects = 13.75, 95% CI [7.39 to 22.24] — Proportion of subjects with severe visual loss was estimated on an observed case basis. Percentage denominator = total number of subjects in the FAS. 95% confidence intervals were calculated from Fleiss quadratic equations

6. Secondary Outcome: Number of Subjects With a Distance Visual Acuity of > 20/200 at Baseline and Progressing to (<= 20/200)
Description: Subjects with improving scores are those with > 20/200 at Baseline and progressing to =< 20/200 at Week 54.
  Subjects with no change are those with > 20/200 at Baseline and remaining at > 20/200 at Week 54.
Time Frame: 54 weeks
Population: FAS; n=77 (number of Subjects at Baseline with >20/200 Visual Acuity)
Measure: Number; unit: participants
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
participants
  Improved | 20
  No Change | 57
Statistical Analysis 1: Comparison: Pegaptanib Sodium; Test type: Superiority or Other; percentage of subjects = 25.97, 95% CI [16.28 to 34.81] — Proportion of subjects progressing to <=20/200 was estimated on an observed case basis. Percentage denominator = total number of subjects in the FAS. 95% confidence intervals were calculated from Fleiss quadratic equations

7. Secondary Outcome: Change in Vision-related Functioning and Quality of Life Using the National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ 25).
Description: Patient reported vision-related functioning and quality of life as measured using the 25 item NEI-VFQ 25. Change = Mean score at 54 weeks - mean score at baseline. A positive change represents an increase in function/health from Baseline. Items grouped as the following - Composite: mean score items 1-25; General Health: item 1; General Vision: item 2; Ocular Pain:4,19; Near Vision:5,6,7; Distance Vision:8,9,14; Social Functioning:11,13; Mental Health Activities:3,21,22,25; Role Difficulties:17,18; Dependency:20,23,24; Driving:15c,16, 16a; Color Vision: 12; Peripheral Vision: 10.
Time Frame: Baseline, 54 weeks or at early termination
Population: FAS; n=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Pegaptanib Sodium
Number analyzed (Participants) | 80
score on scale
  Composite (n=25) | -2.25 (15.71)
  General Health (n=42) | -4.17 (14.52)
  General Vision (n=41) | 3.90 (16.26)
  Ocular Pain (n=43) | 0.35 (15.29)
  Near Vision Activities (n=43) | -3.88 (27.60)
  Distance Vision Activities (n=43) | -6.78 (23.68)
  Social Functioning (n=43) | -0.58 (24.84)
  Mental Health Activities (n=43) | -0.30 (20.45)
  Role Difficulties (n=41) | -4.39 (26.46)
  Dependency (n=41) | -5.28 (22.15)
  Driving (n=27) | -3.70 (30.67)
  Color Vision (n=41) | -1.83 (18.87)
  Peripheral Vision (n=42) | -4.17 (25.25)

ADVERSE EVENTS:
Arm/Group | Pegaptanib Sodium
Serious Adverse Events (participants affected / at risk) | 8
Other Adverse Events (participants affected / at risk) | 28
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Pegaptanib Sodium
Cardiac failure (Cardiac disorders) | 1/81
Cardiac failure acute (Cardiac disorders) | 1/81
Cataract operation (Eye disorders) | 1/81
Macular degeneration (Eye disorders) | 1/81
Peritonitis (Gastrointestinal disorders) | 1/81
Pyelonephritis (Infections and infestations) | 1/81
Angina unstable (Cardiac disorders) | 1/81
Retinal haemorrhage (Eye disorders) | 1/81
Suicide attempt (Psychiatric disorders) | 1/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Pegaptanib Sodium
Conjunctival haemorrhage (Eye disorders) | 6/81
Eye pain (Eye disorders) | 7/81
Macular degeneration (Eye disorders) | 8/81
Myodesopsia (Eye disorders) | 12/81
Pain (General disorders) | 5/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.